CLINICAL TRIAL: NCT04607239
Title: HOme telemonitoRing of Arterial hypertensiOn With antihypertenSive Treatment Titration: a Randomized COntrolled prosPEctive Trial
Brief Title: The Impact of Telemonitoring in the Management of Hypertension
Acronym: HOROSCOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Les Laboratoires des Médicaments Stériles (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HTA-TELEMED
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-10

CONDITIONS: Health Services Administration; Telemedicine; Hypertension
Keywords: Telecommunication; Telecare; Teleconsult; Telemanagement; Telemonitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The interventional group (Telemonitoring) in addition to the usual care group (conventional) will benefit from:
  * a weekly telephone call for collection of home Blood Pressure measurements , therapeutic education & treatment compliance check
  * a monthly call for treatment titration and side effects check
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring (Experimental): In addition to the usual care, this group benefits from a weekly telephone call by the Clinical Research Associate (CRA) for the collection of home blood pressure measurements (which the patient measures twice a day everyday), for therapeutic education, and for treatment compliance assessment.
  This group will also benefit from a monthly call by the attending physician for treatment titration and side effects check.
  Interventions: Procedure: Telemonitoring
- Conventional (Other): This group will benefit form the usual care without any phone calls for therapeutic education, treatment compliance assessment, treatment titration or side effects check.
  The usual care includes attending the follow up visits after inclusion at Day 90 (D-90) & Day 180 (D-180) for face to face consultation with the attending physician.
  Interventions: Procedure: Usual Care without Telemonitoring

INTERVENTIONS:
Procedure: Telemonitoring — * A weekly telephone call by the CRA for the collection of home blood pressure measurements (which the patient measures twice a day everyday), for therapeutic education, and for treatment compliance assessment.
  * A monthly call by the attending physician for treatment titration and side effects check.
  Arms: Telemonitoring
Procedure: Usual Care without Telemonitoring — * Attending the follow up visits after inclusion at Day 90 (D-90) & Day 180 (D-180) for face to face consultation with the attending physician.
  * Usual care without any phone calls for therapeutic education, treatment compliance assessment, treatment titration or side effects check.
  Arms: Conventional

SUMMARY:
Rater blinded, multi-center, prospective, randomized controlled study comparing mean 24 hour systolic blood pressure of eligible hypertensive patients in the TELEMONITORIN group versus the USUAL CARE group, at 6 months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

Included are patients with:

* age ≥ 35 years old
* newly diagnosed hypertention
* uncontrolled hypertention

Exclusion Criteria:

Excluded are patients with:

* orthostatic hypotension
* chronic renal failure (serum creatinine > 200 micromol / L)
* acute coronary syndrome
* coronary revascularization or stroke within the past 3 months
* known secondary causes of hypertension
* pregnancy
* New York Heart Association Class III or IV heart failure or left ventricular ejection fraction < 30%
* dementia or another cause that prevents the application of remote monitoring

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2020-07-04 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Mean of 24h systolic blood pressure (SBP) | 0 - 180 days
  The change from baseline of mean 24-hour systolic blood pressure (SBP) at 6 months of follow-up

SECONDARY OUTCOMES:
Mean of 24h diastolic blood pressure (DBP) | 0-180 days
  The change from baseline of mean 24 hour diastolic blood pressure (DBP) at 6 months of follow-up
percentage of blood pressure load | 0-180 days
  The change of blood pressure load's percentages between baseline and 6 months of follow-up
percentage of Dipping | 0-180 days
  The change of dipping percentages between baseline and 6 months of follow-up
Mean of the Short Form survey (SF-12) scores | 0-180 days
  The change in the mean of SF-12 scores between baseline and 6 months of follow-up
frequency of cardiovascular complications | 180 days
  Clinical outcomes including hospitalization rate, emergency room admissions related to high blood pressure, adverse effects, or other reasons

CONTACTS AND LOCATIONS:
Locations (1):
- Fattouma Bourguiba Hospital, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ben Hafaiedh S, Ben Daya Y, Radoui AH, Bouchoucha M, Razgallah R, Nouira S. Home Telemonitoring of Arterial Hypertension With Antihypertensive Treatment Titration: Protocol for a Randomized Controlled Prospective Trial (HOROSCOPE Study). JMIR Res Protoc. 2022 Mar 1;11(3):e26184. doi: 10.2196/26184. PMID 35230254